CLINICAL TRIAL: NCT05816876
Title: Comparison of Respiratory and Peripheral Muscle Functions, Exercise Capacity and Physical Activity Level in Primary Ciliary Dyskinesia and Kartagener Syndrome
Brief Title: Muscle Function, Exercise Capacity and Physical Activity Level in Primary Ciliary Dyskinesia and Kartagener Syndrome
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof. Dr., Gazi University
Other Study IDs: Gazi University 32
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Primary Ciliary Dyskinesia
Keywords: primary ciliary dyskinesia; exercise capacity; muscle strength; physical activity
MeSH Terms: conditions — Ciliary Motility Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with primary ciliary dyskinesia: Exercise capacity assessed using six minute walk test, physical activity using multi-sensor activity monitor, pulmonary function using spirometry, respiratory muscle strength using mouth pressure device, peripheral muscle strength using hand held dynamometer, respiratory muscle endurance using incremental threshold loading test, life quality using "The Primary Ciliary Dyskinesia Quality of Life scale" (Turkish version).
- Patients with Kartagener Syndrome: Exercise capacity assessed using six minute walk test, physical activity using multi-sensor activity monitor, pulmonary function using spirometry, respiratory muscle strength using mouth pressure device, peripheral muscle strength using hand held dynamometer, respiratory muscle endurance using incremental threshold loading test, life quality using "The Primary Ciliary Dyskinesia Quality of Life scale" (Turkish version).
- Healthy controls: Exercise capacity assessed using six minute walk test, physical activity using multi-sensor activity monitor, pulmonary function using spirometry, respiratory muscle strength using mouth pressure device, peripheral muscle strength using hand held dynamometer, respiratory muscle endurance using incremental threshold loading test, life quality using "The Primary Ciliary Dyskinesia Quality of Life scale" (Turkish version).

SUMMARY:
Studies evaluating respiratory and peripheral muscle functions in PCD patients and comparing them with healthy children are limited in the literature. There is no study investigating pulmonary and extrapulmonary effects in Kartagener syndrome, which is a form of PCD. The aim of our study is to compare respiratory functions, respiratory muscle strength and endurance, exercise capacity, peripheral muscle strength, physical activity level and quality of life in patients with PCD, Kartagener syndrome and healthy children.

DETAILED DESCRIPTION:
Primary ciliary dyskinesia (PCD) is an autosomal recessive disease characterized by abnormal ciliary movement and impaired mucociliary clearance. Kartagener syndrome is an autosomal recessive primary ciliary dyskinesia syndrome characterized by situs inversus, bronchiectasis and chronic sinusitis and is the most serious form of PCD, accounting for 50% of all PCD cases. In these syndromes, there is both movement and structural defect in the cilia, and mucociliary clearance is impaired. Symptoms usually appear in childhood. Organ anomalies can also be seen in Kartagener syndrome. Primary ciliary dyskinesia is a disease that threatens lung functions starting from preschool age. One of the main causes of respiratory muscle weakness in chronic lung diseases is worsening of lung functions. Evaluation of exercise capacity in patients with PCD has prognostic importance. Decreased exercise capacity, respiratory function, and cardiopulmonary function cause physical inactivity. In chronic lung diseases, sedentary lifestyle, airway obstruction, malnutrition and decreased exercise capacity cause muscle weakness. Muscle strength and function are important for performing activities of daily living. There is no study in the literature comparing respiratory and physical functions in children with PCD and in children with Kartagener's syndrome, which is the most serious form of PCD. The aim of our study is to compare respiratory functions, respiratory muscle strength and endurance, exercise capacity, peripheral muscle strength, physical activity level and quality of life in patients with PCD, Kartagener syndrome and healthy children.

The study was planned as a cross-sectional, retrospective. Individuals aged 6-18 years, who were diagnosed with PCD and Kartagener syndrome, and received standard medical treatment, were included in the study. For the healthy group, individuals aged 6-18 years without a known chronic disease were included. Individuals' exercise capacity, respiratory functions, physical activity levels, peripheral and respiratory muscle strength, respiratory muscle endurance and quality of life will be evaluated. Exercise capacity evaluated using six-minute walk test, physical activity using multi-sensor activity monitor, pulmonary function using spirometry, respiratory muscle strength using mouth pressure device, peripheral muscle strength using hand-held dynamometer, respiratory muscle endurance using incremental threshold loading test, life quality using "The Primary Ciliary Dyskinesia Quality of Life scale" (Turkish version). The assessments will be completed in two days.

ELIGIBILITY:
Inclusion Criteria:

Patients;

* Individuals aged 6-18 years, who were diagnosed with PCD and Kartagener syndrome, and received standard medical treatment, were included in the study.

Healthy controls;

-Individuals between the ages of 6 and 18 without a known chronic disease will be included.

Exclusion Criteria:

Patients;

* Patients who are uncooperative, have orthopedic or neurological disorders that will affect functional capacity, and have pneumonia or any acute infection during the evaluation will be excluded from the study.

Healthy controls;

-Those with a known chronic disease, uncooperative and orthopedic or neurological disorders that will affect functional capacity will not be included.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Forty patients with primary ciliary dyskinesia/Kartagener's Syndrome were recruited. It also has 60 healthy data.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Functional exercise capacity | First Day
  Functional exercise capacity will be evaluated with the 6- Minute Walk Test. 6- Minute Walk Test will be applied according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.

SECONDARY OUTCOMES:
Physical activity (Total energy expenditure) | Second Day
  Physical activity was evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient was informed about removing the device while taking a bath. Total energy expenditure (joule / day) was measured with the multi-sensor physical activity monitor. The parameters measured over two days were averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Active energy expenditure (joule / day)) | Second Day
  Physical activity was evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient was informed about removing the device while taking a bath. Active energy expenditure (joule / day) was measured with the multi-sensor physical activity monitor. The parameters measured over two days were averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Physical activity time (min / day)) | Second Day
  Physical activity was evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient was informed about removing the device while taking a bath. Physical activity time (min / day) was measured with the multi-sensor physical activity monitor. The parameters measured over two days were averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Average metabolic equivalent (MET / day)) | Second Day
  Physical activity was evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient was informed about removing the device while taking a bath. Average metabolic equivalent (MET / day) was measured with the multi-sensor physical activity monitor. The parameters measured over two days were averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Number of steps (steps / day)) | Second Day
  Physical activity was evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient was informed about removing the device while taking a bath. Number of steps (steps / day) was measured with the multi-sensor physical activity monitor. The parameters measured over two days were averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Time spent lying down (min / day) days)) | Second Day
  Physical activity was evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient was informed about removing the device while taking a bath. Time spent lying down (min / day) days) was measured with the multi-sensor physical activity monitor. The parameters measured over two days were averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Sleep time (min / day)) | Second Day
  Physical activity was evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient wore the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient was informed about removing the device while taking a bath. Sleep time (min / day) was measured with the multi-sensor physical activity monitor. The parameters measured over two days were averaged and analyzed with the "SenseWear® 7.0 Software" program.
Pulmonary function (Forced vital capacity (FVC)) | First Day
  Pulmonary function was evaluated with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, forced vital capacity (FVC) was evaluated.
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | First Day
  Pulmonary function was evaluated with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, forced expiratory volume in the first second (FEV1) was evaluated.
Pulmonary function (FEV1 / FVC) | First Day
  Pulmonary function was evaluated with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, FEV1 / FVC was evaluated.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | First Day
  Pulmonary function was evaluated with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, flow rate 25-75% of forced expiratory volume (FEF 25-75%) was evaluated.
Pulmonary function (Peak flow rate (PEF)) | First Day
  Pulmonary function was evaluated with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, peak flow rate (PEF) was evaluated.
Respiratory muscle strength | First Day
  Maximal inspiratory (MIP) and maximal expiratory (MEP) pressures expressing respiratory muscle strength were measured with a portable mouth pressure measuring device according to ATS and ERS criteria.
Peripheral muscle strength | Second day
  Isometric peripheral muscle strength was measured with a portable hand dynamometer (JTECH Commander, USA). Measurements were repeated on the shoulder abductors and knee extensors three times on the right and left.
Respiratory muscle endurance | Second Day
  Respiratory muscle endurance was assessed by the POWERbreathe Wellness (POWERbreathe, Inspiratory Muscle Training (IMT) Technologies Ltd., Birmingham, UK) device and the respiratory muscle endurance test at increased threshold load. The test was started with 20% of the maximal inspiratory pressure and the pressure was increased to 40%, 60%, 80% and 100% every two minutes. Patients were asked to continue breathing through the device during the test. During the test, the number of breaths delivered and the maximal time reached during each 2-minute period were recorded. If the individual could not breathe 3 consecutive times, the test was terminated by the physiotherapist. The total duration of the test and the maximum pressure value at which it continues to breathe for at least 1 minute was multiplied. The value found was recorded as the respiratory muscle endurance value.
Life quality | Second Day
  It was evaluated with the Turkish version of the disease-specific Primary Ciliary Dyskinesia Quality of Life scale. The questions were about physical function, emotional function, social function, respiratory symptoms, treatment burden, ear and hearing, sinus symptoms, role function, health perceptions, school functioning, eating and weight problems.

CONTACTS AND LOCATIONS:
Overall Officials: Meral Boşnak Güçlü, Prof. Dr., Study Director — Gazi University; Merve Fırat, MD, Study Chair — Hacettepe University; Şeyma Mutlu, MD, Principal Investigator — Baskent University; Betül Yoleri, MD, Principal Investigator — Gazi University
Locations (1):
- Gazi University Facutly of Health Sciences Department of Physiotheraphy and Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hogg C. Primary ciliary dyskinesia: when to suspect the diagnosis and how to confirm it. Paediatr Respir Rev. 2009 Jun;10(2):44-50. doi: 10.1016/j.prrv.2008.10.001. Epub 2009 Apr 9. PMID 19410200
- [Background] Ortega HA, Vega Nde A, Santos BQ, Maia GT. Primary ciliary dyskinesia: considerations regarding six cases of Kartagener syndrome. J Bras Pneumol. 2007 Sep-Oct;33(5):602-8. doi: 10.1590/s1806-37132007000500017. English, Portuguese. PMID 18026660
- [Background] Takeuchi K, Kitano M, Ishinaga H, Kobayashi M, Ogawa S, Nakatani K, Masuda S, Nagao M, Fujisawa T. Recent advances in primary ciliary dyskinesia. Auris Nasus Larynx. 2016 Jun;43(3):229-36. doi: 10.1016/j.anl.2015.09.012. Epub 2015 Oct 31. PMID 26527516
- [Background] Marthin JK, Petersen N, Skovgaard LT, Nielsen KG. Lung function in patients with primary ciliary dyskinesia: a cross-sectional and 3-decade longitudinal study. Am J Respir Crit Care Med. 2010 Jun 1;181(11):1262-8. doi: 10.1164/rccm.200811-1731OC. Epub 2010 Feb 18. PMID 20167855
- [Background] Arikan H, Yatar I, Calik-Kutukcu E, Aribas Z, Saglam M, Vardar-Yagli N, Savci S, Inal-Ince D, Ozcelik U, Kiper N. A comparison of respiratory and peripheral muscle strength, functional exercise capacity, activities of daily living and physical fitness in patients with cystic fibrosis and healthy subjects. Res Dev Disabil. 2015 Oct-Nov;45-46:147-56. doi: 10.1016/j.ridd.2015.07.020. Epub 2015 Aug 1. PMID 26241869
- [Background] Firat M, Bosnak-Guclu M, Sismanlar-Eyuboglu T, Tana-Aslan A. Respiratory muscle strength, exercise capacity and physical activity in patients with primary ciliary dyskinesia: A cross-sectional study. Respir Med. 2022 Jan;191:106719. doi: 10.1016/j.rmed.2021.106719. Epub 2021 Dec 17. PMID 34952415
- [Background] Simsek S, Inal-Ince D, Cakmak A, Emiralioglu N, Calik-Kutukcu E, Saglam M, Vardar-Yagli N, Ozcelik HU, Sonbahar-Ulu H, Bozdemir-Ozel C, Kiper N, Arikan H. Reduced anaerobic and aerobic performance in children with primary ciliary dyskinesia. Eur J Pediatr. 2018 May;177(5):765-773. doi: 10.1007/s00431-018-3121-2. Epub 2018 Feb 27. PMID 29487997
- [Background] Denizoglu Kulli H, Gurses HN, Zeren M, Ucgun H, Cakir E. Do pulmonary and extrapulmonary features differ among cystic fibrosis, primary ciliary dyskinesia, and healthy children? Pediatr Pulmonol. 2020 Nov;55(11):3067-3073. doi: 10.1002/ppul.25052. Epub 2020 Sep 11. PMID 32877003
- [Background] Madsen A, Green K, Buchvald F, Hanel B, Nielsen KG. Aerobic fitness in children and young adults with primary ciliary dyskinesia. PLoS One. 2013 Aug 19;8(8):e71409. doi: 10.1371/journal.pone.0071409. eCollection 2013. PMID 23977038